CLINICAL TRIAL: NCT05747729
Title: A Single-arm, Open-label, Single-center Clinical Trial of Surufatinib and Serplulimab Combined With Standard Chemotherapy (Platinum/Etoposide) in Neuroendocrine Carcinoma.
Brief Title: A Single-arm, Open-label, Clinical Trial of Surufatinib/Serplulimab/Platinum/Etoposide in Neuroendocrine Carcinoma.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIONEC
Record Dates: First submitted 2023-02-18; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib/Serplulimab/Platinum/Etoposide (Experimental)
  Interventions: Drug: Surufatinib and Serplulimab

INTERVENTIONS:
Drug: Surufatinib and Serplulimab — Surufatinib: Safety lead-in : Oral, QD, starting dose 250 mg, adjusted according to DLT. Dose expansion: administration according to the dose determined in the safety lead-in phase.
  Serplulimab: 300 mg intravenous infusion on day 1, repeated every 3 weeks.

SUMMARY:
This study is a prospective open-label, single-arm, single-center clinical study. Patients with neuroendocrine carcinoma who had not previously received standard therapy were enrolled in this study once they have signed the informed consent form (ICF) and been identified as eligible in screening. This clinical trial evaluates the efficacy and safety of surufatinib and serplulimab combined with standard chemotherapy (Platinum/Etoposide) in neuroendocrine carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. With histologically or cytologically confirmed extra-pulmonary neuroendocrine carcinoma (including mixed neuroendocrine or non-neuroendocrine tumors [at least 30% neuroendocrine carcinoma component]);
3. Previously untreated with systemic therapy;
4. age ≥18 years;
5. Have at least one measurable lesion according to RECIST v1.1;
6. ECOG performance status: 0-1;
7. Expected survival time > 3 months;
8. For evidence of sufficient organ functions, the subjects shall meet the following laboratory parameters: 1) Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without use of granulocyte colony stimulating factor in recent 14 days; 2) Platelet count ≥ 100 × 109/L without blood transfusion in recent 14 days; 3) Hemoglobin > 9 g/dL without blood transfusion or erythropoietin use in recent 14 days; 4) Total bilirubin ≤ 1.5 × upper limit of normal (ULN); or total bilirubin > ULN, direct bilirubin ≤ ULN; 5) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (ALT or AST ≤ 5 × ULN for patients with liver metastasis); 6) Blood creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by Cockcroft- Gault formula) ≥ 50 mL/min;
9. Women of childbearing potential need to use at least one medically approved contraceptive measure (such as intrauterine device, contraceptive pill or condom) during the study treatment and within 180 days after the end of the study treatment; Before the first dose, serum HCG examination must be negative; and women must be non-lactating.

Exclusion Criteria:

1. Neuroendocrine carcinoma of the lung;
2. With known allergic reactions to the drugs in this study;
3. Unable or unwilling to swallow Surufatinib or suffering from significant digestive system diseases that may interfere with absorption, metabolism, or excretion;
4. With clinically significant or uncontrolled heart diseases, including unstable angina, acute myocardial infarction within 6 months before the first dose, grade III/IV congestive heart failure (New York Heart Association), and uncontrolled arrhythmia (subjects with pacemakers or with atrial fibrillation but well controlled heart rate are allowed); With ECG changes or medical history considered clinically significant by the investigator; QTc interval > 450 ms for male or > 470 ms for female at screening;
5. With active ulcers, intestinal perforation, and intestinal obstruction;
6. With active bleeding or bleeding tendency;
7. With uncontrolled hypertension (systolic pressure > 150 mmHg or diastolic pressure > 100 mmHg) after the optimal medical treatment;
8. Urine protein ≥ ++ and the amount of urine protein in 24 hours >1.0g;
9. Any active autoimmune disease requiring systemic treatment or with a history of autoimmune disease within 2 years, including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, hypophysitis, vasculitis, systemic lupus erythematosus, etc. (Vitiligo, psoriasis, alopecia or Grave's disease without systemic treatment within the past 2 years, and type I diabetic patients who only need insulin replacement therapy can be included); with a history of primary immunodeficiency; patients only with positive autoimmune antibody need to confirm according to the investigator;
10. Received systemic immunostimulant therapy within 4 weeks before the first dose;
11. Received any live vaccines or live attenuated vaccines within 4 weeks prior to the first dose or planned to be administered live vaccines or live attenuated vaccines during the study;
12. Pleural effusion, ascites, or pericardial effusion with obvious clinical symptoms that require drainage;
13. Diagnosed with malignant tumors within 5 years before the first dose, excluding radically cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ;
14. Presence of severe infection in the active phase or with poor clinical control;

    1. With known history of human immunodeficiency virus (HIV) infection or confirmed with positive immune test results;
    2. Acute or chronic active hepatitis B or C infection; hepatitis B virus (HBV) DNA > 2000 IU/mL or 104 copies/mL; hepatitis C virus (HCV) RNA > 103 copies/mL; or other hepatitis, liver cirrhosis.
15. Symptomatic brain metastases (confirmed or suspected)
16. The investigator confirms that the patients has any clinical or laboratory abnormalities who are not suitable for participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 7 years
  Progression-Free Survival (PFS) According to RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China